CLINICAL TRIAL: NCT01456663
Title: A Single-dose, Open-label, Parallel Study to Assess the Pharmacokinetics of AFQ056 in Subjects With Mild, Moderate and Severe Hepatic Impairment Compared to Healthy Control Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics of AFQ056 in Subjects With Hepatic Impairment Compared to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CAFQ056A2123; 2011-000748-28 (EudraCT Number)
Record Dates: First submitted 2011-08-24; First posted 2011-10-21 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2013-02

CONDITIONS: Hepatic Impairment
Keywords: AFQ056; Hepatic impairment; Hepatic impaired
MeSH Terms: interventions — mavoglurant

ARMS (1):
- AFQ056 (Experimental)
  Interventions: Drug: AFQ056

INTERVENTIONS:
Drug: AFQ056

SUMMARY:
This study will assess the pharmacokinetics of AFQ056 in subjects with mild, moderate, severe hepatic impairment compared with healthy control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Groups 1, 2, 3 and 4 (all subjects)
* Male and female Caucasian subjects
* Group 1, 2 and 3 (subjects with hepatic impairment)
* Subjects must satisfy the criteria for hepatic impairment as evidenced by a Child-Pugh score of A, B or C at screening
* Group 4 (healthy subjects)
* Each healthy subject must match in age (±8 years), gender, weight (±15%) to an individual subject with hepatic impairment in group 1, 2 or 3.

Exclusion Criteria:

* Groups 1, 2, 3 and 4 (all subjects)
* Use of any tobacco products from 1 week prior to cotinine screening assessments until study completion.
* Group 1, 2 and 3 (subjects with hepatic impairment)
* History of drug or alcohol abuse within 3 months prior to screening
* History or presence of any clinically significant disease of any major system organ class including (but not limited to) cardiovascular, metabolic, renal, neurological or psychiatric diseases within 1 month prior to study drug administration except for hepatic impairment or any other disease associated with this underlying condition.
* Any surgical or medical condition other than hepatic impairment which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the safety of the study subject in case of participation in the study.
* History or presence of encephalopathy within 6 months prior screening (except for subjects in Groups 2 and 3).
* Documented presence of a porto-systemic shunt.
* Documented presence of esophagus varices (stage III or IV).
* Group 4 (healthy subjects)
* History or presence of any clinically significant disease of any major system organ class including (but not limited to) cardiovascular, metabolic, renal, neurological or psychiatric diseases.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the safety of the study subject in case of participation in the study. History of drug or alcohol abuse within 12 months prior to screening, or evidence of such abuse as indicated by the laboratory assays conducted during screening and baseline.
* History or presence of hepatitis B or C and/or positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result at screening.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2011-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Measure: Profile of Pharmacokinetics of AFQ056 in each subjects groups | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 12, 24, 36, 48, 72, 96, 120 hours post-dose
  AUClast, AUCinf, Cmax, Tmax, T1/2, CL/F, Vz/F

SECONDARY OUTCOMES:
Measure: : Number of subjects with adverse event in each group | From dose administration (day 1) to 13+/- 2 days after the single dose administration
  Number and type of adverse events, number and type of findings in standard laboratory results, special laboratory results (Hypothaliamic-pituitary axis, porphyrin profile) electrocardiogram holters, or in vital signs
Measure: Plasma protein binding results of AFQ056 in each groups. | 2 hours after single dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Novartis Investigative Site, Orlando, Florida, United States
- Novartis Investigative Site, Berlin, Germany
- Novartis Investigative Site, Balatonfüred, Hungary

REFERENCES:
- See also: Results for CAFQ056A2123 can be found on the Novartis Clinical Trial Results website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=9464